CLINICAL TRIAL: NCT04612348
Title: Utility of POC Gastric Ultrasound in Confirming Stomach is Empty in Intubated Patients Fed Gastrically (NG) Versus Transpylorically (NJ) to Ensure Low Risk of Aspiration.
Brief Title: Gastric Ultrasound in Tube Fed Intubated Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chair, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: STUDY00001377
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- NJ tube fed: Critically ill children receiving nutrition via a nasojejunal feeding tube.
  Interventions: Diagnostic Test: Ultrasound
- NG tube fed: Critically ill children receiving nutrition via a nasogastric feeding tube.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Point of care ultrasound to measure gastric contents.

SUMMARY:
This study will use point of care (POC) gastric ultrasound to confirm that nasojejunal tube (NJ) feeds result in minimal to no gastric content and therefore are low risk for aspiration and should be allowed at the very least to decrease the time that enteral feeds need to be held prior to a procedure or if they need to be held at all. This would allow critically ill children to receive the nutrition that they need to heal for longer periods of time. Using ultrasound would also potentially eliminate the need for exposure to x-rays to confirm tube placement. Most ICUs have a POC ultrasound machine so this would be any easy tool to access to improve patient care.

ELIGIBILITY:
Inclusion Criteria:

* all PICU patients intubated < 7 days that are receiving NJ or NG feeds

Exclusion Criteria:

* patients that cannot be moved
* patients with significant GI conditions affecting motility
* patients intubated for more than seven days

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Critically ill children at Nationwide Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastric contents | Baseline (Day 1)
  Amount of gastric contents measured by ultrasound.

SECONDARY OUTCOMES:
Gastric contents | Day 2 (if still intubated & being tube fed)
  Amount of gastric contents measured by ultrasound.
Gastric contents | Day 3 (if still intubated & being tube fed)
  Amount of gastric contents measured by ultrasound.
Gastric contents | Day 4 (if still intubated & being tube fed)
  Amount of gastric contents measured by ultrasound.
Gastric contents | Day 5 (if still intubated & being tube fed)
  Amount of gastric contents measured by ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Tobias, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States